CLINICAL TRIAL: NCT05155215
Title: A Phase 1-2 Study to Evaluate the Safety and Efficacy of IM19 CAR-T Cells in Patients With Relapsed and Refractory (R/R) Mantle Cell Lymphoma
Brief Title: Study to Evaluate the Safety and Efficacy of IM19 CAR-T Cells in Patients With Relapsed and Refractory (R/R) Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SD46
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Lymphoma; Lymphoma, Mantle-Cell; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM19 CAR-T cells (Experimental)
  Interventions: Biological: IM19 CAR-T cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: IM19 CAR-T cells — IM19 CAR-T cells will be administered at dose level: 100×10^6 CAR-T cells or 200×10^6 CAR-T cells
Drug: Cyclophosphamide — 300 mg/m^2 per day for 3 days (IV)
Drug: Fludarabine — 30 mg/m^2 per day for 3 days (IV)

SUMMARY:
This is a phase I/II, open-label, multicenter study to assess the efficacy and safety of IM19 CAR-T cells in adult R/R Mantle Cell Lymphoma subjects

ELIGIBILITY:
Inclusion Criteria:

* Subjects with relapsed or refractory mantle cell lymphoma, diagnosed as CD19 positive by cytology or histology；
* Subjects have measurable positive lesion according to Lugano Classification;
* ≥ 18 years old;
* Expected survival is greater than 3 months；
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* The toxicity caused by the previous treatment has stabilized or recovered to ≤1 level (except for the case where the investigator judges that it has no clinical significance);
* Women of childbearing age who had a negative blood pregnancy test before the start of the trial and agreed to take effective contraceptive measures during the trial period until the last follow-up; male subjects with fertility partners agreed to take effective contraceptive measures during the trial period until the last follow-up;
* Adequate organ function;
* Adequate vascular access for leukapheresis procedure;
* Volunteer to participate in this trial and sign on the informed consent.

Exclusion Criteria:

* Central nervous system (CNS) involvement by lymphoma;
* Received allo-hematopoietic stem cell transplantation or organ transplantation therapy previously；
* Subjects with cardiac atrial or cardiac ventricular lymphoma involvement；
* Serous effusion with symptoms of compression;
* History of autoimmune disease (eg Crohn's disease, rheumatoid arthritis, systemic lupus) within the last 2 years;
* Presence of acute or chronic graft-versus-host disease (GVHD);
* Use prohibited drugs or treatments within a specified period of time before cell collection；
* Received anti-CD19 target therapy (unless the CD19 target test is still positive);
* Received CAR-T cell therapy;
* Received the study drug within 4 weeks before cell collection. However, if the trial treatment is invalid or the disease progresses, and at least 5 half-lives have passed before the cell collection, it is allowed to enter the group;
* Received radiotherapy within 6 weeks prior to cell collection, including large bone marrow areas such as the sternum or pelvis. Subjects who have progressed in the radiotherapy site or have PET-positive lesions in other non-irradiated sites are eligible to be included in the group;
* Received donor lymphocyte infusion (DLI) within 6 weeks before CAR-T cell infusion;
* If anti-PD1, PD-L1 and other immunotherapies have been used before CAR-T cell reinfusion, at least 5 half-lives must elapse between the last medication and before CAR-T cell reinfusion;
* History or presence of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, cerebral edema, posteriorreversible encephalopathy syndrome, or any autoimmune disease with CNS involvement;
* Received autologous transplantation within 6 weeks before the start of screening;
* Subjects has HBV, HCV, HIV ,EBV,ECV or syphilis infection at the time of screening;
* Live vaccine received within 6 weeks before the start of screening;
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina,active arrhythmias, or other clinically significant cardiac disease within 6 months of enrollment;
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment;
* History of malignancy other than nonmelanomatous skin cancer or carcinoma in situ (eg, cervix, bladder, breast) unless disease-free for at least 3 years；
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management. Simple urinary tract infection (UTI) and bacterial pharyngitis are permitted if the investigator evaluates that it can be controlled by treatment, they can be included in the group;
* In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and abnormal laboratory test results as assessed by CTCAE V5.0 | Up to 28 days after IM19 CAR-T cell infusion
Objective response rate (ORR) | At 3 months after IM19 CAR-T cell infusion
  ORR, defined as the proportion of participants with a complete response or partial response, as determined by the investigator according to Lugano(2014)

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 28 days and 6 months after IM19 CAR-T cell infusion
  ORR, defined as the proportion of participants with a complete response or partial response, as determined by the investigator according to Lugano(2014)
Progression-free survival (PFS) | Up to 24 weeks after IM19 CAR-T cell infusion
  PFS, defined as the time from CAR-T cell infusion to the first occurrence of disease progression or death from any cause (whichever occurs first) , as determined by the investigator according to Lugano(2014)
Duration of Response (DOR) | Up to 24 weeks after IM19 CAR-T cell infusion
  DOR, defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first) in Stage 1, as determined by the investigator according to Lugano(2014)
Overall survival (OS) | Up to 24 weeks after CAR-T cell infusion
  OS , defined as the time from IM19 CAR-T cell infusion to death from any cause
Persistence of CAR-T cells (cell counts and cell percentage in peripheral blood) | Up to 24 weeks after IM19 CAR-T cell infusion
  The persistence over time of CAR T cells in the peripheral blood as determined by flow cytometry and qPCR
Anti-therapeutic IM19 CAR-T cells antibody | Up to 24 weeks after IM19 CAR-T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Jing, Ph.D, Principal Investigator — Peking University Third Hospital